CLINICAL TRIAL: NCT06197321
Title: Non-invasive Prediction of Fluid and Noradrenaline Responsiveness in Critical Care Patients Using the Carotid Wave Intensity (cWI)
Brief Title: Non-invasive Prediction of Fluid and Noradrenaline Responsiveness Using the Carotid Wave Intensity.
Acronym: VACC
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Frederique de Raat, Principal Investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: nWMO-2023.131
Record Dates: First submitted 2023-12-05; First posted 2024-01-09 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-09

CONDITIONS: Shock; Aortic Valve Disease; Coronary Artery Disease; Mitral Valve Disease
Keywords: Ventriculo-arterial coupling; Carotid ultrasound
MeSH Terms: conditions — Shock; Aortic Valve Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to study a new method to compute ventricular-arterial coupling (VAC) in adult intensive care patients after cardiac surgery. VAC is a metric that describes the interaction between the heart and the arterial system. The new method of measuring VAC uses carotid ultrasound measurements. The main questions this study aims to answer are:

* Can VAC measured using carotid ultrasound predict the hemodynamic response to drugs?
* What is the concordance of VAC measurements obtained via carotid ultrasound with VAC measurements obtained via the standard, single-beat method? Measurements will be performed in the operating room and at the ICU.

DETAILED DESCRIPTION:
The goal of this prospective observational study is to study ventricular-arterial coupling (VAC) measured using carotid ultrasound in adult intensive care patients after cardiac surgery. The objectives of this study are:

* To determine if VAC measured using carotid ultrasound can predict the hemodynamic response to drugs.
* To assess and quantify the concordance of VAC measurements obtained using carotid ultrasound with VAC measurements obtained using the single-beat method.

Measurements will be performed in the operating room and at the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Admitted to the ICU after cardiac surgery

Exclusion Criteria:

* No informed consent for study participation
* Within the first 3 hours of ICU admission noradrenaline infusion is not increased or started, and/or a fluid bolus is not given; both on indication of the attending physician
* Patient with chronic obstructive pulmonary disease (COPD) gold stage 3 or 4
* Pregnancy
* Moderate to severe aortic valve disease
* Atrial fibrillation
* Carotid artery stenosis >50%
* History of cerebrovascular accident or transient ischemic attack
* History of cerebral trauma
* Morbid obesity (BMI >40 kg/m2)
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients after cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The prediction of the hemodynamic response to norepinephrine or fluids using carotid ultrasound measurements. | Through study completion, an average of 1 year.
  It will be studied if carotid ultrasound measurements can be used to predict a hemodynamic response to hemodynamic drugs, where the hemodynamic response is defined as a 15% increase in stroke volume.

SECONDARY OUTCOMES:
The concordance of ventricular-arterial coupling (VAC) measurements obtained using carotid ultrasound measurements with VAC measurements obtained using the single-beat method. | Through study completion, an average of 1 year.
  The concordance between VAC measurements obtained using carotid ultrasound and VAC measurements obtained using the single-beat method will be assessed and quantified.

CONTACTS AND LOCATIONS:
Overall Officials: R. A. Bouwman, Prof., Study Chair — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No